CLINICAL TRIAL: NCT05977764
Title: Role of Contrast-enhanced Ultrasound (CEUS) and Shear Wave Elastography (SWE) to Characterize Focal Liver Lesions (FLLs)
Brief Title: Multimodal Ultrasound and Focal Liver Lesions (FLLs)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2824
Record Dates: First submitted 2023-03-16; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lesion target (Experimental): CEUS on lesion target
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Contrast enhanced ultrasound

SUMMARY:
Background and aim: FLLs are common findings in abdominal ultrasound and differential diagnosis between benign and malignant lesions is often challenging, especially in patients with chronic liver diseases. The diagnostic role of CEUS has already been defined by international guidelines when lesions show a typical pattern for hepatocellular carcinoma whereas in case of non-typical contrast enhanced patterns radiologic imaging or liver biopsy are still needed. However, these techniques are more invasive and expensive than ultrasound. Therefore, the aim of this study is to identify D-CEUS and SWE quantitative parameters useful for characterizing FLLs.

Study design: Prospective, observational, single-center study Methods: 50 consecutive adult patients with focal liver lesions detectable with B-mode ultrasound will be enrolled in the Unit of Internal Medicine and Gastroenterology of the Policlinico Gemelli. Exclusion criteria will be liver failure, hearth failure, previous locoregional or systemic treatments for FLLs (e.g. ablation, chemoembolization, alcoholization, chemotherapy), known allergy to ultrasound contrast agents. After obtaining informed consent and identifying the target lesion in B-mode ultrasound, patients will undergo CEUS and SWE and, subsequently, to computed tomography/magnetic resonance/biopsy according to international guidelines and current clinical practice. The average, maximum, minimum and standard deviation value of lesion elasticity in KPa will be calculated using SWE. Three consecutive SWE acquisitions will be performed both for the lesion and for the liver parenchyma and the average value of the three measurements will be considered. The CEUS will allow the construction of signal intensity curves as a function of time in a specific area of interest drawn manually. From these curves a series of quantitative parameters related to the flow and volume of blood will be extrapolated and in particular: peak intensity, PI (in Arbitrary Units, AU); time to peak, TP ( in seconds); area under the time curve, AUC (in AU); slope of the wash-in curve, Pw (in AU per second); average transit time, MTT (in seconds). In addition, the personal, clinical and laboratory data necessary to determine the hepatological scores of disease severity such as MELD and Child-Pugh will be collected. The study has an expected duration of one year.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* adult patients (more than 18 years old)
* focal liver lesions detectable with B-mode ultrasound

Exclusion Criteria:

* liver failure,
* hearth failure,
* previous locoregional or systemic treatments for FLLs (e.g. ablation, chemoembolization, alcoholization, chemotherapy),
* known allergy to ultrasound contrast agents
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
to identify D-CEUS quantitative parameters useful for characterizing FLLs. | one month after liver biopsy
  to quantify peak enhancement intensity, PI (in Arbitrary Units, AU), measured by analysing D-CEUS time-intensity curves, in patients with FLLs undergoing liver biopsy and stratified according to the histologic exam.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Assunta Zocco, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy